CLINICAL TRIAL: NCT02223195
Title: Biomarkers in Saliva in Children With Juvenil Idiopathic Arthritis
Status: Completed | Type: Observational
Sponsor: Folktandvården Stockholms län AB (Other Government)
Responsible Party: Principal Investigator, Malin Collin, PhD student, DDS, Folktandvården Stockholms län AB
Other Study IDs: MC 2
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile Idiopathic Arthritis; Saliva
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva sampels
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose and aims This as a pilot study that aims to investigate which inflammatory biomarkers can be found in saliva in children with Juvenile Idiopathic Arthritis (JIA).

The hypothesis is that children with JIA will show a different pattern of inflammatory biomarkers in saliva than healthy Children.

The null hypothesis is that there are no differences.

DETAILED DESCRIPTION:
This is a comparison between 100 children with JIA and 100 healthy children. Saliva will be collected and analyzed with respect to biomarkers.

One-hundred consecutive patients with active JIA, as diagnosed by the Department of Pediatric Rheumatology, Astrid Lindgrens Barnsjukhus, Karolinska University Hospital will be included.

Inclusion criteria are:

* age between 7 and 14 years
* a diagnosis of JIA according to the International League of Associations for rheumatology

Exclusion criteria are:

* current malignancies
* TMJ surgery or trauma within two years
* recent intra-articular glucocorticoid injection in TMJ (within 1 month)
* other conditions or diseases than JIA that may cause orofacial pain. The parents of the patients and/or the patients will give their verbal and written informed consent to participate in the study according to the permission from the regional ethical committee 2011/2:1.

The control group of 100 age and sex matched healthy children will be included at Folktandvården Stockholms Län AB.

Inclusion criteria are:

• age between 7 and 14 years

Exclusion criteria are:

* current malignancies
* TMJ surgery or trauma within two years
* recent intra-articular glucocorticoid injection in TMJ (within 1 month)
* A diagnosis of JIA
* other conditions or diseases than JIA that may cause orofacial pain. The parents of the patients and/or the patients will give their verbal and written informed consent to participate in the study according to the permission from the regional ethical committee 2011/2:1.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of JIA according to the International League of Associations for rheumatology (ILAR) The parents of the patients and/or the patients will give their verbal and written informed consent to participate in the study according to the permission from the regional ethical committee 2011/2:1

Exclusion Criteria:

1. current malignancies
2. TMJ surgery or trauma within two years
3. Recent intra-articular glucocorticoid injection in TMJ (within 1 month)
4. Other conditions or diseases than JIA that may cause orofacial pain. Fore the controllgroup JIA are excluded

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Group 1: 40 consecutive patients with active JIA, as diagnosed by the Department of Pediatric Rheumatology, Astrid Lindgrens Barnsjukhus, Karolinska University Hospital will be included.
  Group 2: 40 healthy children, age-and sex-matched.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Biomarkers in saliva, a comparison between healthy children and children with juvenile idiopathic arthritis. | one day
  Saliva sampels will be colleceted and analysed

CONTACTS AND LOCATIONS:
Overall Officials: Britt Hedenberg Magnusson, PhD DDS, Principal Investigator — Karolinska Institutet
Locations (1):
- Folktandvården Stockholmslän AB, Stockholm, Sweden